CLINICAL TRIAL: NCT04519307
Title: Evaluation of Newborns Presenting With Suspected COVID 19: A Single Center Experience
Brief Title: Evaluation of Newborns Presenting With Suspected COVID 19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Senem Alkan Özdemir, Associate Professor of Neonatology, Dr. Behcet Uz Children's Hospital
Other Study IDs: 2020/251
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Viral Infection
Keywords: newborn; covid infection; viral infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The newborns with covid 19 infection
- Group 2: The newborns with no covid 19 infection

SUMMARY:
This study evaluates the newborns who had respiratory symptoms at the neonatal intensive care admission

ELIGIBILITY:
Inclusion Criteria:

* All newborns who had respiratory symptoms at the NICU admission

Exclusion Criteria:

* Congenital abnormalities

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns who had respiratory symptoms at the NICU admission
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
General Characteristics of the infants with respiratory infection at the NICU admission | 5 months
  Demographical characteristics will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Dr. Behcet Uz Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes